CLINICAL TRIAL: NCT01763125
Title: Establishment of a Blood Sample Bank in the Field of Gynaecological Oncology.
Brief Title: Establishment of a Tumor Bank for Blood Samples
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Robert Zeillinger, Dr.phil., Prof. Dr., Medical University of Vienna
Other Study IDs: EK 366/2003
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Neoplasms of the Female Genitalia; Lung Neoplasms; Endocrine Gland Neoplasms
Keywords: circulating tumor cells; CTC; tumor marker
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Endocrine Gland Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Universal tumor bank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Malignant tumors: Patients who have one of the Neoplasms stated above under "conditions". Blood samples will be taken.
  Interventions: Other: Blood collection
- Benign controls: Patients with a benign tumor or an inflammatory disease - to be matched by age and affected organ with a patient with a malignant disease.
  Blood samples will be taken.
  Interventions: Other: Blood collection
- Healthy controls: People/patients who have no known disease at time of blood sampling or are admitted to the hospital for minor interventions and have no inflammatory disease.
  Blood samples will be taken.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood sample is collected during routine blood collection by a medical doctor. No more than 60ml (max.) at one timepoint.

SUMMARY:
Establishment of a tumor bank, consisting of blood samples of tumor patients and healthy people as controls. The blood samples will be collected systematically together with the corresponding clinical data. The biological samples, the clinical date together with prospective experimental date constitute the entity of the tumor bank.

DETAILED DESCRIPTION:
Recent progress in diagnosis and therapy of cancer diseases can be ascribed mainly to translational research. The relevance of "translational oncology" will only increase in the future -"From bench to bedside" - the swift implementation of new science research results in clinical studies in order to expedite progress in clinical cancer therapy for the benefit of the patient.

Its almost a matter of course in the medical science today to collect biological samples together with clinical information thereby creating the foundation for future excellent fundamental research.

The aim of this tumor bank is to consist of biological samples (together with a tissue bank - see EK 260/2003) and isolates of tumor patients and healthy people as controls. The biological samples, the clinical date together with prospective experimental date constitute the entity of the tumor bank. The content of the tumor bank can provide essential material for current and future research (e.g. analyses of prognostic or predictive tumor markers; genetically analysis (polymorphism, mutation, hypermethylation; verification and characterisation of disseminated tumor cells).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* Age 18 to 90 years max.
* Just one current known malignant disease or
* Just one current inflammatory disease

Exclusion Criteria:

* Inflammatory disease and malignant disease
* multiple malignancies
* multiple diseases
* underage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Male and female patients/people.
  * Minimum age 18 years
  * Characteristics: Recruited at the Medical University Vienna or at one of the facilities cooperating with the Vienna Med. University
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2003-11; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Establishment of blood/tissue bank consisting of oncological samples from cancer patients and benign and healthy controls. | 14 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeillinger, Prof.Dr., Principal Investigator — Medical University Vienna, Dept. of Obstetrics & Gynaecology
Locations (6):
- Innsbruck Medical University, Innsbruck, Austria
- University Hospitals Leuven - Department of Obstetrics and Gynaecology, Leuven, Belgium
- Germany (3):
  - Charité University - Campus Virchow Chlinic, Berlin
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Clinic of Ruhr University Bochum, Herne
- European Institute of Oncology, Division of Gynecologic Oncology, Unit of Preventive Gynecology, Milan, Italy

REFERENCES:
- [Result] Hefler LA, Concin N, Hofstetter G, Marth C, Mustea A, Sehouli J, Zeillinger R, Leipold H, Lass H, Grimm C, Tempfer CB, Reinthaller A. Serum C-reactive protein as independent prognostic variable in patients with ovarian cancer. Clin Cancer Res. 2008 Feb 1;14(3):710-4. doi: 10.1158/1078-0432.CCR-07-1044. PMID 18245530
- [Result] Konigsberg R, Gneist M, Jahn-Kuch D, Pfeiler G, Hager G, Hudec M, Dittrich C, Zeillinger R. Circulating tumor cells in metastatic colorectal cancer: efficacy and feasibility of different enrichment methods. Cancer Lett. 2010 Jul 1;293(1):117-23. doi: 10.1016/j.canlet.2010.01.003. Epub 2010 Feb 18. PMID 20167419
- [Result] Obermayr E, Sanchez-Cabo F, Tea MK, Singer CF, Krainer M, Fischer MB, Sehouli J, Reinthaller A, Horvat R, Heinze G, Tong D, Zeillinger R. Assessment of a six gene panel for the molecular detection of circulating tumor cells in the blood of female cancer patients. BMC Cancer. 2010 Dec 3;10:666. doi: 10.1186/1471-2407-10-666. PMID 21129172
- [Result] Konigsberg R, Obermayr E, Bises G, Pfeiler G, Gneist M, Wrba F, de Santis M, Zeillinger R, Hudec M, Dittrich C. Detection of EpCAM positive and negative circulating tumor cells in metastatic breast cancer patients. Acta Oncol. 2011 Jun;50(5):700-10. doi: 10.3109/0284186X.2010.549151. Epub 2011 Jan 24. PMID 21261508
- [Result] Obermayr E, Castillo-Tong DC, Pils D, Speiser P, Braicu I, Van Gorp T, Mahner S, Sehouli J, Vergote I, Zeillinger R. Molecular characterization of circulating tumor cells in patients with ovarian cancer improves their prognostic significance -- a study of the OVCAD consortium. Gynecol Oncol. 2013 Jan;128(1):15-21. doi: 10.1016/j.ygyno.2012.09.021. Epub 2012 Sep 24. PMID 23017820
- [Derived] Hasenburg A, Eichkorn D, Vosshagen F, Obermayr E, Geroldinger A, Zeillinger R, Bossart M. Biomarker-based early detection of epithelial ovarian cancer based on a five-protein signature in patient's plasma - a prospective trial. BMC Cancer. 2021 Sep 16;21(1):1037. doi: 10.1186/s12885-021-08682-y. PMID 34530759